CLINICAL TRIAL: NCT01316848
Title: A Phase 1, Single Center, Open-label, Randomized, Two-period Crossover Food Effect Study of Single Doses of Tivozanib (AV-951) in Healthy Subjects
Brief Title: A Single Center, Open-label, Randomized, Two-period Crossover Food Effect Study of Single Doses of Tivozanib (AV-951) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-10-115
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Food Effect of Tivozanib in Health Subjects
Keywords: AV-951; tivozanib; healthy Subjects; food Effect; pharmacokinetics
MeSH Terms: interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted dosing followed by fed dosing (Experimental): Dosing in the fasted state followed by fed dosing
  Interventions: Drug: tivozanib
- Fed dosing followed by fasted dosing (Experimental): Dosing in the fed state followed by fasted dosing
  Interventions: Drug: tivozanib

INTERVENTIONS:
Drug: tivozanib — tivozanib 1.5 mg capsule, 2 discrete single doses separated by 6-weeks
  Other Names: AV-951

SUMMARY:
This study will determine the effect of food on the pharmacokinetics (PK) of a single dose of 1.5 mg tivozanib in normal healthy subjects.

DETAILED DESCRIPTION:
This study will be an open-label, randomized, two-period, crossover PK food effect study of tivozanib administered orally at 1.5 mg. Subjects will be screened for eligibility up to 28 days prior to entry into the study.

For each of 2 study periods, subjects will be admitted to the clinical research unit (CRU) on the day before dosing and fast overnight (approximately 10 hours). On the morning of dosing for each of the 2 study periods, subjects will receive a single oral dose of 1.5 mg tivozanib in either the fasted or fed state. Subjects will remain at the CRU for at least 48 hours after administration of study drug for collection of serial blood samples for pharmacokinetic (PK) analysis and safety monitoring. Subjects will return to the CRU on an outpatient basis for collection of additional blood samples for up to 504 hours postdose.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, between 18 and 55 years of age, inclusive.
* Body mass index (BMI) within the range of 18.5 to 31.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs.
* Clinical laboratory evaluations (including a chemistry panel comprised of 20 analytes [Chem-20; fasted at least 10 hours], complete blood count [CBC], and urinalysis [UA] not exceeding 2 x ULN or less than 2 x LLN, unless deemed not clinically significant by the Investigator.
* Nonsmokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to Screening), verified by a cotinine test at Screening and each study period Check-in.
* Negative test for selected drugs of abuse at Screening (does not include alcohol) and at each study period Check-in (does include alcohol; Appendix A).
* Negative hepatitis panel (including hepatitis B virus surface antigen [HBsAg] and hepatitis C virus antibody [anti-HCV] and negative human immunodeficiency virus(HIV) antibody screens (Appendix A).
* Females who are not pregnant, non-lactating, and either postmenopausal for at least 1 year, surgically sterile (eg, tubal ligation, hysterectomy, etc.) for at least 90 days prior to screening, or agree to use at least one of the following forms of contraception from informed consent until 45 days after Study Completion: a non-hormonal intrauterine device with spermicide; female condom with spermicide; contraceptive sponge with spermicide; diaphragm with spermicide; cervical cap with spermicide; a male sexual partner who agrees to use a male condom with spermicide; or a sterile sexual partner; For all females, a serum pregnancy test result must be negative at Screening and each study period Check-in.
* Male subjects who are either sterile or agree to use, during the period from informed consent until 45 days following Study Completion, 1 of the following approved methods of contraception: a double barrier method (eg, male condom with spermicide, use by female sexual partner of an intrauterine device with spermicide, a female condom with spermicide, contraceptive sponge with spermicide, a diaphragm with spermicide, or use of a cervical cap with spermicide); a sterile sexual partner; a female sexual partner using an intravaginal system (eg,NuvaRing®); or a partner using an oral, implantable, transdermal, or injectable contraceptives.
* Able to comprehend and willing to sign an informed consent form (ICF).

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic/endocrine, allergic, dermatological, hepatic, renal, hematological, pulmonary, immune, cardiovascular, gastrointestinal, genitourinary, neurological, or psychiatric disorder(as determined by the Investigator).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
* History of stomach or intestinal surgery, nephrectomy, cholecystectomy or resection that would potentially alter absorption and/or excretion of orally administered drugs as determined by the investigator (appendectomy and/or hernia repair may be allowed).
* History or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant.
* Diagnosis of alcoholism or drug addiction within 1 year prior to Period 1 Check-in.
* Participation in any other investigational drug study in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer prior to informed consent.
* Use of any prescription medications or products within 14 days prior to Period 1 prior to informed consent.
* Use of any over-the-counter (OTC), non-prescription preparations (including vitamins, minerals, and phytotherapeutic, herbal, dietary supplements, or plant derived preparations) within 7 days prior to each study period Check-in.
* Use of alcohol-, grapefruit-, Seville orange-, or caffeine-containing foods, juices, or beverages within 72 hours prior to each study period Check-in.
* Use of known hepatic or renal clearance altering agents (eg, erythromycin, cimetidine, barbiturates, phenothiazines, or herbal/plant derived preparations such as St. John's Wort, etc.) for a period of 60 days prior to informed consent;
* Poor peripheral venous access.
* Donation of blood ≥ 250 mL from 30 days prior to informed consent until study completion, inclusive, or of plasma from 2 weeks prior to informed consent until study completion, inclusive.
* Receipt of blood products within 2 months prior to Period 1 Check-in;
* Blood pressure greater than 140/90 mmHg confirmed by repeat at Screening or at Period 1 Check-in.
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the effect of food on the PK of a single dose of 1.5 mg tivozanib in normal healthy subjects. | Planned Enrollment/Screening Duration: Approximately 4 weeks. Length of Each Confinement: Approximately 24 hours prior to dose until approximately 48 hours postdose. Planned Study Conduct Duration: Approximately 13 weeks
  Blood samples for PK analysis of serum tivozanib levels will be collected for a 3-week period following each of 2 doses.

SECONDARY OUTCOMES:
To assess the safety and tolerability of single doses of 1.5 mg tivozanib. | Planned Enrollment/Screening Duration: Approximately 4 weeks. Length of Each Confinement: Approximately 24 hours prior to dose until approximately 48 hours postdose. Planned Study Conduct Duration: Approximately 13 weeks
  Safety will be assessed by physical exam, clinical laboratory evaluations and ECGs.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A. King, MD, Principal Investigator — Covance Clinical Research Unit - Dallas
Locations (1):
- Covance Clinical Research Unit, Inc., Dallas, Texas, United States